CLINICAL TRIAL: NCT01924429
Title: Neurobiological Basis of Response to Vyvanse in Adults With ADHD: an fMRI Study of Brain Activation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jeffrey Newcorn (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Newcorn, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GCO 09-1186
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: ADHD
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; fMRI; Imaging; Vyvanse; Stimulant Medication; Treatment; Clinical Trial; Adult
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- On Drug then off Drug (Experimental): Participants receive fMRI #1 on drug, #2 off drug Escalating stepped titration: 30, 50 or 70mg
  Interventions: Drug: Lisdexamfetamine
- Off drug then on drug (Experimental): Participants receive fMRI #1 off drug, #2 on drug Escalating stepped dose titration: 30, 50, 70mg
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine — Escalating stepped dose titration: 30, 50 or 70mg
  Other Names: Vyvanse

SUMMARY:
The purpose of this study is to determine the effects of Vyvanse, an FDA approved medication used in the treatment of Attention Deficit Hyperactivity Disorder (ADHD), on brain activity in adults with attention-deficit hyperactivity disorder (ADHD). Participants may qualify for participation in this study because they have ADHD and are willing to participate in two Functional Magnetic Resonance Imaging (fMRI) scans and receive Vyvanse for treatment of their symptoms. Another purpose of this study is to collect and bank samples of blood for research to examine how genes influence brain activation seen during the brain scans. The study also seeks to find out whether certain genes are related to ADHD. Participants' entire genetic makeup will not be determined from this sample.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV-TR diagnosis of adult ADHD (inattentive, hyperactive-impulsive or combined subtype), established via the ACDS v1.2.
* Must be between 18-55 years, inclusive.
* Provides written informed consent.

Exclusion Criteria:

* Lifetime or current diagnosis of bipolar disorder, schizophrenia or schizoaffective disorder.
* Current diagnosis of comorbid major depressive disorder, anxiety disorder or dysthymia or any controlled (i.e. requires pharmacological treatment) comorbid diagnosis. Participants with uncontrolled depressive or anxiety disorders may participate if, in the opinion of the Principal Investigator, the disorder will not confound the results of efficacy or safety assessments, increase risk to the participant or lead to difficulty complying with the protocol.
* Meets current DSM-IV-TR criteria for alcohol or any non-alcohol substance abuse or dependence disorder.
* Have organic brain disease (such as dementia) or traumatic brain injury residua. Have a history of seizure disorder (other than febrile seizures) or participants who have taken (or are currently taking) anticonvulsants for seizure control.
* Females who are currently pregnant or breast feeding, and women of child-bearing potential who are not currently using an adequate form of birth control.
* Participants with clinically significant abnormalities in ECG results that are deemed exclusionary in the opinion of the Principal Investigator will not be allowed in the trial.
* Participants who work the night shift or another schedule that would preclude beginning the daily dose of study medication in the morning.
* Participants with a positive urine drug result at Screening.
* Medical conditions limiting participation in the study.
* Documented history of intolerance or non-responsivity to methylphenidate or amphetamines.
* Have a medical condition that would, in the opinion of the study physician, make participation medically hazardous.
* ADHD, Not Otherwise Specified
* History of surgery involving metal implants, metal fragments in the eyes, braces, or a pacemaker.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Newcorn JH, Ivanov I, Krone B, Li X, Duhoux S, White S, Schulz KP, Bedard AV, Pedraza J, Adler L, Blair RJ. Neurobiological basis of reinforcement-based decision making in adults with ADHD treated with lisdexamfetamine dimesylate: Preliminary findings and implications for mechanisms influencing clinical improvement. J Psychiatr Res. 2024 Feb;170:19-26. doi: 10.1016/j.jpsychires.2023.11.037. Epub 2023 Dec 3. PMID 38101205
- [Derived] Schulz KP, Krone B, Adler LA, Bedard AV, Duhoux S, Pedraza J, Mahagabin S, Newcorn JH. Lisdexamfetamine Targets Amygdala Mechanisms That Bias Cognitive Control in Attention-Deficit/Hyperactivity Disorder. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Aug;3(8):686-693. doi: 10.1016/j.bpsc.2018.03.004. Epub 2018 Mar 19. PMID 29661516

RESULTS

PARTICIPANT FLOW:
Groups:
- On Drug Then Off Drug: Participants receive fMRI #1 on drug, #2 off drug Escalating stepped titration: 30, 50 or 70mg
  Lisdexamphetamine: Escalating stepped dose titration: 30, 50 or 70mg
- Off Drug Then on Drug: Participants receive fMRI #1 off drug, #2 on drug Escalating stepped dose titration: 30, 50, 70mg
  Lisdexamphetamine: Escalating stepped dose titration: 30, 50 or 70mg
Period: Period 1 - First Intervention (4 Weeks)
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Started | 17 | 13
Completed | 17 | 13
Not Completed | 0 | 0
Period: Washout Period (2 Weeks)
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Started | 17 | 13
Completed | 14 | 11
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: Period 2 - Second Intervention (4 Weeks)
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- On Drug, Then Off Drug: fMRI #1 on drug, #2 off drug
- Off Drug, Then on Drug: fMRI #1 off drug, #2 on drug
- Total: Total of all reporting groups
Arm/Group | On Drug, Then Off Drug | Off Drug, Then on Drug | Total
Number analyzed (Participants) | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.46 (11.82) | 37.27 (11.81) | 35.84 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Go/No-Go Task Percentage Assessed by fMRI
Description: Performance Measures on the Go/No-Go Task assessed by fMRI as a Function of Trial Type, Face Emotion, and Drug Condition in Adults with Attention-Deficit/Hyperactivity Disorder. The Go/No-Go Task is a neuropsychological test that provides a direct measure of number of responses made that are "correct" or "incorrect". It is not a scale. Reported are the percentage of correct responses on that direct performance measure. 0% correct is worse than 100% correct.
Time Frame: 8 weeks
Population: Performance measures are done while participants are off drug and while on drug.
Measure: Mean (Standard Error); unit: percentage correct responses/inhibitions
Groups:
- Placebo: Participants received fMRI while off drug
- Lisdexamfetamine: Participants received fMRI while on drug
Arm/Group | Placebo | Lisdexamfetamine
Number analyzed (Participants) | 25 | 25
percentage correct responses/inhibitions
  Happy Correct Responses | 91.7 (2.8) | 97.0 (3.8)
  Happy Correct Inhibitions | 88.7 (9.4) | 87.9 (11.5)
  Sad Correct Responses | 90.3 (7.7) | 88.5 (10.6)
  Sad Correct Inhibitions | 84.4 (12.5) | 86.7 (11.3)
  Neutral Correct Responses | 93.2 (12.2) | 95.6 (5.8)
  Neutral Correct Inhibitions | 77.5 (12.3) | 79.6 (11.6)

2. Primary Outcome: fMRI Reaction Time
Description: Reaction-time, as measured by the reaction time test Go/No-Go Task as a Function of Trial Type, Face Emotion, and Drug Condition in Adults with Attention-Deficit/Hyperactivity Disorder
Time Frame: up to 6 weeks
Measure: Mean (Standard Error); unit: ms
Arm/Group | Placebo | Lisdexamfetamine
Number analyzed (Participants) | 25 | 25
ms
  Happy | 532 (99) | 519 (114)
  Sad | 533 (110) | 509 (96)
  Neutral | 553 (109) | 533 (104)

3. Secondary Outcome: BRIEF-A
Description: Behavior Rating Inventory of Executive Function®-Adult Version (BRIEF-A): Norm Referenced Measure of Impaired Executive Functioning, reported in T-Scores (0 to 100, with 50 +/-1 SD = 'Normal', higher is worse, more impaired)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 14 | 11
t-score | 66.64 (11.89) | 73.5 (14.75)

4. Secondary Outcome: BRIEF-A
Description: Behavior Rating Inventory of Executive Function®-Adult Version (BRIEF-A): Norm Referenced Measure of Impaired Executive Functioning, reported in T-Scores (higher is worse)
Time Frame: at one week
Population: not collected
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: BRIEF-A
Description: as for outcome 4
Time Frame: at 4 weeks
Population: not collected
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: ASRS - Expanded
Description: ADHD and Related Symptoms Measure (ASRS): self report, reported as Sum of Responses (0-4 per item, higher = more impaired) 0-26 (normal range) and >27 (clinically significant symptoms).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 14 | 11
units on a scale | 83.7 (25.59) | 86 (4.24)

7. Secondary Outcome: ASRS - Expanded
Description: as for outcome 6
Time Frame: at one week
Population: not collected
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: ASRS - Expanded
Description: as for outcome 6
Time Frame: at 4 weeks
Population: not collected
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: WRAADS
Description: The Wender-Reimherr adult attention deficit disorder scale (WRAADS): Symptom measure for emotional functioning/lability, generally reported as Sum of Responses (0-2 per item, higher = more impaired).
  For this outcome measure, Average scores for particular questions were taken - specifically question 3, question 4, and question 5.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 14 | 11
units on a scale
  Question 3 | 0.80 (0.86) | 0.94 (0.745)
  Question 4 | 1.27 (1.22) | 1.47 (1.23)
  Question 5 | 1.13 (1.35) | 1.82 (1.19)

10. Secondary Outcome: ADHD-RS-IV Combined Sum
Description: ADHD symptoms and severity. Norm referenced interview to assess severity and frequency of ADHD symptoms. 18 Items are scored 0-3 to reflect severity and frequency of ADHD symptoms, and a sum is taken. Full range from 0 to 54, with higher number indicating more symptoms and severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 14 | 11
units on a scale
  On Drug | 11.00 (6.98) | 13.67 (11.64)
  Placebo | 25.65 (8.53) | 31.00 (14.80)

11. Secondary Outcome: ADHD-Inattentive
Description: ADHD symptoms and severity - subscale for Inattentiveness. 9-item scale, each scored 0-3, with total from 0 to 27. Higher score indicates higher level of inattentiveness.
Time Frame: 4 weeks and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 14 | 11
units on a scale
  On drug | 7.36 (4.53) | 8.83 (7.63)
  Placebo | 18.94 (6.21) | 19.2 (5.07)

12. Secondary Outcome: CGI-I
Description: Clinical Global Impressions - CGI-I: Clinical response was the Clinical Global Impression-Improvement scale (CGI-I). Lower CGI-I scores indicate greater improvement (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 14 | 11
units on a scale | 1.88 (1.13) | 2.00 (1.41)

13. Secondary Outcome: CGI-S
Description: CGI-S: Severity of impairment due to ADHD was measured by the Clinical Global Impressions-Severity scale (CGI-S). Lower scores indicate less severe impairment from symptoms, with a CGI-I=1 indicating the person is "normal" with no impairment. (1= normal, not ill, 2= minimally ill, 3= mildly ill, 4= moderately ill, 5=markedly ill, 6=severely ill, 7= very severely ill)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Drug Then Off Drug | Off Drug Then on Drug
Number analyzed (Participants) | 14 | 11
units on a scale | 4.9 (1.0) | 4.95 (0.9)

ADVERSE EVENTS:
Groups:
- On Drug, Then Off Drug: Participants receive fMRI #1 on drug, #2 off drug Escalating stepped titration: 30, 50 or 70mg
  Lisdexamphetamine: Escalating stepped dose titration: 30, 50 or 70mg
- Off Drug, Then on Drug: Participants receive fMRI #1 off drug, #2 on drug Escalating stepped dose titration: 30, 50, 70mg
  Lisdexamphetamine: Escalating stepped dose titration: 30, 50 or 70mg
Arm/Group | On Drug, Then Off Drug | Off Drug, Then on Drug
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 14/14 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | On Drug, Then Off Drug (N=14) | Off Drug, Then on Drug (N=11)
Incidental finding on brain scan (General disorders) | 0 | 1 — benign
Incidental Physical finding (General disorders) | 3 | 0 — benign
Insomnia (General disorders) | 2 | 1
Heart Racing (General disorders) | 1 | 0 — secondary to anxiety
Dry mouth (General disorders) | 1 | 2
feeling agitated (General disorders) | 1 | 0 — counseled to reduce caffeine
Tired (General disorders) | 1 | 0
Anxious (General disorders) | 1 | 2
Headache (General disorders) | 1 | 2
Restless (General disorders) | 1 | 0
Seasonal allergies (General disorders) | 0 | 2
Subjectively feeling "stuck" (General disorders) | 0 | 1 — no motivation
Suspiciousness (General disorders) | 1 | 0
Backache (Musculoskeletal and connective tissue disorders) | 1 | 0
Reduced Appetite (General disorders) | 1 | 0
Skin Sores (Skin and subcutaneous tissue disorders) | 1 | 0
Bruxism (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No